CLINICAL TRIAL: NCT05267210
Title: Turkish Translation, Cultural Adaptation, Validity and Reliability Study of the Back Pain and Body Posture Assessment Questionnaire
Brief Title: Turkish Translation, Validity and Reliability of the Back Pain and Body Posture Assessment Questionnaire
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, Ayşenur Gökşen, PhD, Karamanoğlu Mehmetbey University
Other Study IDs: 07-2021/38
Record Dates: First submitted 2022-02-23; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — 1. Back Pain and Body Posture Assessment Instrument for Adults (BackPDE-Y) This questionnaire assesses pain and risk factors associated with back pain. The questionnaire includes questions that include demographic, socio-economic, hereditary and behavioral risk factors. The questionarie consists of 20 questions in total.
  2. Musculoskeletal Health Questionnaire (CIS-SS) The questionnaire included pain/stiffness (during the day and night), physical function (walking and dressing), physical activity level, involvement of symptom-related work/daily life and social activities/hobbies, difficulty sleeping, fatigue, emotional well-being, diagnosis and It consists of a total of 14 questions evaluating the understanding of the treatment and the overall effect of the disease.

SUMMARY:
The Adult Back Pain and Body Posture Assessment Instrument (BackPDE-Y), whose validity and reliability is planned, will be applied. This assessment scale will be translated into Turkish by two native Turkish speakers, one who is fluent in English.

DETAILED DESCRIPTION:
220 people aged between 20-65 are planned to be included in the study. The data obtained from the study will be analyzed with appropriate statistical methods.

In addition, a previously valid and reliable Musculoskeletal System Health Inquiry (MIS-SS) questionnaire, which evaluates the musculoskeletal problems of individuals included in the Study, will be applied. It will be evaluated whether the results of the data obtained from the Back Pain and Body Posture Assessment Instrument for Adults (BackPDE-Y), which we have validated in Turkish, and the results of the data obtained from the Musculoskeletal Health Questionnaire (CIS-SS) questionnaire are consistent with each other.

ELIGIBILITY:
Inclusion Criteria:

18-65 years old Willingness to participate in the study The mother tongue is Turkish, Being able to read and write, - It is between the ages of 18-65.

Exclusion Criteria:

Those with a known or concomitant diagnosis of dementia Not wanting to participate in the study Patients with psychotic disorders, depression with psychotic symptoms, bipolar depression Having a psychiatric illness with a serious psychiatric illness that may prevent the individual from understanding and completing the questionnaire

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: According to the power analysis, the number of samples was calculated to be at least 10 times the number of items in the scale. 220 people aged between 18-65 will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Estimated)
Dates: Start 2021-10-02 (Actual); Primary Completion 2022-08-02 (Estimated); Study Completion 2022-09-02 (Estimated)

PRIMARY OUTCOMES:
Back Pain and Body Posture Assessment Instrument for Adults (BackPDE-Y) total score | 6 month
  The total score will be obtained by adding the points obtained from the answers given to the questionnaire.

SECONDARY OUTCOMES:
Musculoskeletal Health Questionnaire (CIS-SS) | 6 month
  The total score will be obtained by adding the points obtained from the answers given to the questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşenur Gökşen, Principal Investigator — Karamanoğlu Mehmetbey University
Locations (1):
- Karamanoglu Mehmetbey University, Karaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erdinc O, Hot K, Ozkaya M. Turkish version of the Cornell Musculoskeletal Discomfort Questionnaire: cross-cultural adaptation and validation. Work. 2011;39(3):251-60. doi: 10.3233/WOR-2011-1173. PMID 21709361